CLINICAL TRIAL: NCT02877550
Title: A Phase I Trial of Obinutuzumab in Combination With Venetoclax in Previously Untreated Follicular Lymphoma Patients
Brief Title: Obinutuzumab in Combination With Venetoclax in Previously Untreated Follicular Lymphoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 35/15; 2017-001175-23 (EudraCT Number)
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Follicular Lymphoma
Keywords: untreated Follicular lymphoma; non-Hodgkin lymphoma; Obinutuzumab; Gazyva; Gazyvaro; Venetoclax; Venclexta
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part A - dose escalation and part B - dose expansion (Experimental): Part A: dose escalation:
  Combination therapy N= 4-18 pts Cycle 1-6 (1 cycle = 28 days) Obinutuzumab: 1000 mg, i.v. infusion; d1, 8, 15 C1 and d1 C2-6 Venetoclax: p.o. once daily according to dose level (DL)
  Part B - dose expansion:
  Combination therapy N= up to 25 pts Cycle 1-6 (1 cycle = 28 days) Obinutuzumab: 1000 mg, i.v. infusion d1, 8, 15 C1 and d1 C2-6 Venetoclax: p.o. once daily according to MTD
  Part A and part B are followed (in case of no PD) by an obinutuzumab maintenance therapy for 2 years
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab: 1000 mg, i.v. infusion; d1, 8, 15 C1 and d1 C2-6
  Other Names: GA101; Gazyvaro; Gazyva
Drug: Venetoclax — p.o. once daily according to dose level (DL) or MTD
  Other Names: ABT-199; GDC-0199; Venclexta

SUMMARY:
Follicular lymphoma (FL) is an indolent yet incurable lymphoma characterized by initial responses to standard therapies, invariably followed by shorter disease free intervals. Obinutuzumab, a novel type II, anti-CD20 monoclonal antibody has been approved in combination with chlorambucil for the treatment of previously untreated chronic lymphocytic leukemia (CLL) and in combination with bendamustine followed by obinutuzumab alone for FL who did not respond to, or who progressed during or after treatment with rituximab or a rituximab-containing regimen, or in relapse after such treatment. Additionally, venetoclax, a small molecule Bcl-2 inhibitor, showed single agent activity in relapsed/refractory (R/R) CLL and other B-cell lymphomas, including R/R FL. Preclinical evidence suggests a synergism of the two drugs in vitro as well as in different lymphoma in vivo models. Based on single agent clinical activity and on the preclinical data of the combination of both drugs and aiming to develop a new chemotherapy-free combination regimen, this trial plans to evaluate the combination of obinutuzumab and venetoclax in previously untreated FL patients in need of systemic therapy. This phase I study will provide information on the safety and tolerability together with evidence of preliminary antitumor activity. Combination treatment consists of a 6 cycles of 28 days each. The combination therapy is followed by a 2 years maintenance with obinutuzumab. Dosing of obinutuzumab is as per Swissmedic approval in FL.Venetoclax will be administered in different dose levels according to the trial design.

DETAILED DESCRIPTION:
Follicular lymphoma is an indolent yet incurable lymphoma characterized by a relapsing-remitting course with initial responses to standard therapies, invariably followed by shorter disease free intervals. In recent years, significant treatment improvements have been achieved, mainly due to the introduction of the anti-CD20 monoclonal antibody rituximab in standard therapies. Unfortunately, most patients invariably relapse and require additional treatment. Therefore new therapies are needed in order to further improve treatment outcomes.

Recent advances in preclinical research and the improved knowledge of the molecular biology of lymphomas have permitted the development of a high number of new therapeutic compounds that inhibit components of altered signaling pathways that drive the genesis of lymphomas and their progression. Additionally, improvements in monoclonal antibody technology have permitted the development of new and active monoclonal antibodies that recognize different antigens on the surface of the lymphoma cells.

Obinutuzumab, a type II, anti-CD20 monoclonal antibody has been clinically tested both as single agent as well as in combination with chemotherapy or targeted agents, showing significant clinical activity in CLL and in FL patients that were refractory to rituximab.

Additionally venetoclax, a small molecule Bcl-2 inhibitor has recently advanced into clinical trials, showing a good safety profile and signs of single agent activity in CLL and other B-cell lymphomas, including patients with relapsed/refractory FL. There is interest to further investigate venetoclax in FL, given that the pathogenesis of this lymphoma relies on the chromosomal translocation t(14;18)(q32;q21), which is present in nearly all cases and results in constitutive overexpression of the BCL2 gene, allowing B cells to abrogate the default germinal center apoptotic program.

The combination of these two compounds is interesting given their single agent activity observed in FL. Preclinical studies have demonstrated a synergism both in vitro as well as in vivo models in different lymphomas and the two compounds are currently investigated in combination studies in CLL and with the chemotherapy CHOP regimen in non-Hodgkin lymphomas.

Based on the single agent activity of the two compounds and aiming to develop a new chemotherapy-free combination regimen, this SAKK trial plans to evaluate the combination of obinutuzumab and venetoclax in previously untreated FL patients in need of systemic therapy. There are data with venetoclax in combination with rituximab and bendamustine in relapsed or refractory Non-Hodgkin lymphoma (NHL) patients. No significant safety signal has been observed.

In the indication CLL the combination of obinutuzumab and venetoclax is currently investigated in a phase I dose finding trial (NCT01685892). In the currently ongoing CLL 14 trial the combination of obinutuzumab plus venetoclax is randomly compared to obinutuzumab plus chlorambucil within a prospective phase III study. Nevertheless, to the best of our knowledge, the proposed trial is one of the first trials worldwide investigating the combination treatment of obinutuzumab with venetoclax in FL as first line treatment. Given the need to further improve chemotherapy-free approaches in the first-line treatment of patients with FL in need of systemic therapy, this combination may provide an opportunity for an active and well tolerated regimen that does not present the short and long term toxicities of chemotherapy.

This phase I study will provide information on the safety and tolerability together with evidence of preliminary antitumor activity of obinutuzumab in combination with venetoclax in the first line treatment of FL.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration.
* Histological diagnosis of FL CD20+; grade 1, 2, 3a; stage III+IV; stage II not suitable for radiotherapy; all FLIPI
* In need of first systemic therapy
* At least one two-dimensionally measurable nodal lesion with a longest diameter (LDi) ˃15 mm or a measurable extra nodal lesion with a LDi ˃ 10 mm in CT, PET/CT scan (preferable) or MRI, according to Cheson et al, 2014
* Bone marrow biopsy within 6 months.
* Age18-80 years
* WHO performance status 0-2
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function
* Women of childbearing potential have a negative serum (beta-human chorionic gonadotropin [β-hCG]) pregnancy test within 3 days before inclusion into the trial.

Exclusion Criteria:

* FL stage I
* Transformation to high-grade DLBCL prior to therapy
* FL grade 3 b
* Indolent lymphoma other than FL
* Known primary central nervous system (CNS) lymphoma
* Known CNS or leptomeningeal involvement
* Previous systemic FL therapies
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Concurrent treatment with other experimental drugs or other anticancer therapy in a clinical trial within 30 days prior to registration.
* Live-virus vaccines treatment within 28 days prior to registration
* Patients regularly taking corticosteroids during the last 30 days, unless administered at a dose equivalent to prednisone ≤ 15 mg/day for indications other than lymphoma or lymphoma-related symptoms
* Women who are breastfeeding
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV), unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), uncontrolled hypertension (sustained systolic blood pressure > 150 mm Hg and/or diastolic > 100 mm Hg despite antihypertensive therapy)
* History of cerebrovascular accident or intracranial hemorrhage within 6 months prior to registration
* Known history of

  * human immunodeficiency virus (HIV)
  * active/chronic Hepatitis C
  * active/chronic Hepatitis B Virus infection (HBsAg+ and/or HBcAb+)
  * or any active systemic infection requiring intravenous (iv) antimicrobial treatment.

Patients with a history of recurring or chronic infections may be included in the study but caution should be exercised and an infectious disease expert should be consulted before enrollment in the trial.

* Requires anticoagulation with vitamin K antagonists (e.g. phenprocoumon, warfarin)
* Coagulation parameters

  * INR ˃1.5x ULN
  * PT or PTT/aPTT ˃1.5x ULN
* Requires treatment with strong CYP3A inhibitors (such as fluconazole, ketoconazole, and clarithromycin) and strong CYP3A inducers (such as rifampin, carbamazepine, phenytoin, St. John's wort) 7 days prior to registration
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information (if applicable) or most recent IB (if approved product information not available)
* Known hypersensitivity to trial drugs or to any component of the trial drugs
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies. Known sensitivity or allergy to murine products
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment, affect patient compliance or place the patient at high risk from treatment-related complications.
* Psychiatric disorder precluding understanding information of trial-related topics, giving informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) during the first cycle | Day 28 of the first cycle
  The primary endpoint is the frequency of DLTs which are relevant for the determination of the maximum tolerated dose (MTD) in the dose escalation phase of the trial.

SECONDARY OUTCOMES:
Adverse events (AEs) | at 6 months (combination therapy) and at 2 years (maintenance therapy)
Laboratory safety variables | at 6 months (combination therapy) and at 2 years (maintenance therapy)
Complete response (CR) | at 6 months and 30 months
Overall response (OR) based on best response observed during combination therapy. | at 6 months, based on best response observed during combination therapy, at 30 months and based on best response observed during whole therapy (combination and maintenance)
Duration of response | at 2.5 years
Progression free survival (PFS) | at 12 months, at 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Stathis, MD, Study Chair — IOSI -Ospedale San Giovanni, Bellinzona
Locations (6):
- Switzerland (6):
  - Universitaetsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital, Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Kantonsspital - St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stathis A, Mey U, Schar S, Hitz F, Pott C, Mach N, Krasniqi F, Novak U, Schmidt C, Hohloch K, Kienle DL, Hess D, Moccia AA, Unterhalt M, Eckhardt K, Hayoz S, Forestieri G, Rossi D, Dirnhofer S, Ceriani L, Sartori G, Bertoni F, Buske C, Zucca E, Hiddemann W. SAKK 35/15: a phase 1 trial of obinutuzumab in combination with venetoclax in patients with previously untreated follicular lymphoma. Blood Adv. 2022 Jul 12;6(13):3911-3920. doi: 10.1182/bloodadvances.2021006520. PMID 35537101